CLINICAL TRIAL: NCT06690008
Title: Comparison of the Effectiveness and Feasibility of Two Fluoride Therapies for Caries Management in Early Childhood: a Randomized Clinical Trial
Brief Title: Fluoride Caries-control Effectiveness/Feasibility in Children
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universidad El Bosque, Bogotá (Other)
Collaborators: Corporacion Universitaria Rafael Nunez (Other); Cooperative University of Colombia (Other)
Responsible Party: Principal Investigator, Stefania Martignon, Principal Investigator, Universidad El Bosque, Bogotá
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: PCI-2022-11045
Record Dates: First submitted 2024-06-25; First posted 2024-11-15 (Actual); Last update posted 2025-04-15 (Actual); Status verified 2025-04

CONDITIONS: Caries,Dental
Keywords: Dental caries; Fluorides; Diamine silver fluoride; Sodium fluoride; Prevention; Control
MeSH Terms: conditions — Dental Caries

STUDY DESIGN:
Intervention Model Description: Participants are assigned to two groups in parallel for the duration of the study
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Experimental group (SDF group) (Experimental): SDF application: -Vaseline will be used to isolate and protect the soft tissues (gums and lips); -Then, SDF will be dispensed on paraffin paper according to the dosage guide; - SDF will be applied on dental surfaces and rubbed with a micro-applicator (1'); -Patients will be asked not to eat/drink/rinse (30').
  Interventions: Procedure: Experimental group
- Control group NaF group) (Active Comparator): NaF application: - NaF will be dispensed according to the dosage guide; -all tooth surfaces will be brushed with NaF; -The patient will close his/her mouth until NaF get hard; -Patients will be asked not to eat/drink/rinse (30') Do not brush teeth that day.
  Interventions: Procedure: Experimental group

INTERVENTIONS:
Procedure: Experimental group — SDF application

SUMMARY:
The aim of this study is to compare the effectiveness and feasibility of using silver diamine fluoride solution (SDF) vs. sodium fluoride varnish (NaF) for caries management in children from Bogotá (and its suburban areas) and Cartagena, in terms of: 1. Preventive effect: number of carious dental surfaces (cavitated); 2. Arrest effect: number of arrested carious tooth surfaces (cavitated); 3. Presence and number of adverse effects in soft/hard oral tissues.

Null hypothesis: Effectiveness and feasibility of silver diamine fluoride is superior to the sodium fluoride for caries management:

Alternative hypothesis: Effectiveness and feasibility of silver diamine fluoride is not superior to the sodium fluoride for caries management.

This Randomize Clinical Trial included 752 3-4 year-old medically healthy children from Bogotá and Cartagena. Participants were randomized equality distributed per city to receive either SDF (38%) or NaF (5%) biannually. Primary outcomes: cavity prevention and arresting effect. Secondary: feasibility (adherence, fidelity), dental-care parental satisfaction/acceptance and adverse effects. Data were analysed using t-tests, Chi-square, and Generalized estimating equations -GEE (0.05 statistical significance).

DETAILED DESCRIPTION:
Ethical approval obtained from the Ethics Board at Universidad El Bosque (UEB 2022-11045).

It corresponds to a double-blind randomised controlled clinical trial following the Consolidated Standards of Reporting and Trials Checklist (CONSORT) 2010.

Population: 3-4-year-old children from (Bogotá and Cartagena) with good self-reported general health.

Sample size was calculated according to the protocols of Gao et al. and Chu et al. [20,21] (using Program-Sample-Size®, version 1.1), considering type-I error: 0.05; type-II error: 0.10; standard deviation: 0.87; expected average group-1: 0.47, group-2: 0.70. The determined sample size was of n=601, increasing due to possible losses by 25% (n=151) for a total sample size of n=752, equally divided in n=376 per arm (Bogotá/Cartagena).

Once the informed consent is signed by the parents, a comprehensive examination will be performed, including:

Ethical approval obtained from the Ethics Board at Universidad El Bosque (UEB 2022-11045).

Randomized, double blind, active controlled Clinical Trial. Population: 3-4-year-old children from (Bogotá and Cartagena) with good self-reported general health.

Sample size Sample size was calculated, according to the protocol of Gao et al. (2021) and Chu et al. (2002) (Program-Size-of-Sample®, version 1.1), considering type-I error: 0.05; type-II error: 0.10; standard deviation: 0.87; expected average group-1: 0.47, group-2: 0.70. Determined sample size: n=601, plus 25% (n=75) (dropout), for a total of: n=752, n=376/arm, evenly split (Bogotá/Cartagena).

Participants: In Cartagena and Bogotá (including surrounding areas), researchers invited children from private daycare centers, kindergartens associated with the Colombian Family Welfare Institute (ICBF), and charities to participate in a study. In 2022, they reached out to leaders of 12 centers in low-socioeconomic-status areas in Cartagena, and in 2022/2023, they contacted leaders of 37 centers in low and lower-middle socioeconomic areas in Bogotá. Ultimately, six centers in Cartagena and 32 in Bogotá agreed to participate, representing around 1,130 children.

On examination days, informed consent was obtained from the parents or guardians of 842 children aged 3-4 years (Cartagena: n=392; Bogotá: n=450). Exclusion criteria included children with systemic diseases, disabilities, regular medication use, unwillingness to participate, or families planning to move within the next year. Recruitment continued until the sample size was met. The study involved baseline and 1-year follow-up dental examinations.

Baseline and 1-year follow-up dental examinations: The dental assessments were conducted in community rooms using portable dental units, headlights, basic instruments (including a round-tip probe), and gauze/cotton rolls for drying. After children received assisted toothbrushing with 1450 ppm fluoride toothpaste, six calibrated examiners assessed caries using ICDAS visual criteria. Inter-examiner reproducibility (weighted Kappa: 0.71-0.80) and intra-examiner reproducibility (weighted Kappa: 0.75-0.92) were achieved.

Caries lesions were classified using the ICDAS-merged Epi criteria, which divides lesions by severity: Initial (non-cavitated, ICDAS 1-2), Moderate (microcavity or underlying shadow, ICDAS 3-4), and Extensive (cavity, ICDAS 5-6). Caries activity was determined through gentle probing: Active (soft or leathery dentine) or Inactive (shiny and hard dentine). Fillings and teeth missing due to caries were also recorded. This assessment was repeated at the 1-year follow-up, with intra-examiner reproducibility confirmed on 10% of assessments (weighted Kappa: 0.73-0.93 initially and 0.76-0.97 at follow-up).

Demographic characteristics and Oral health behaviors: At baseline, using previously established questionnaires, two research assistants conducted interviews with parents or caregivers to gather information on the children's socio-demographic characteristics (age, sex) and oral health-related practices. These included daily toothbrushing frequency, fluoride toothpaste use, daily consumption of free sugars, preventive dental care, and symptomatic-based dental visits.

Randomization: After the dental assessment in each city, children were randomly assigned to one of two intervention groups (NaF or SDF) by the coordinator using opaque, sequentially numbered envelopes in the presence of an external assistant. The randomization process followed the order of each child's arrival and was blind to the examiner. Stratified randomization was done at each site in a 1:1 ratio using Stata 14.0 software (Stata Corp, College Station, Texas USA). The randomization and allocation sequence were independently supervised by one of the authors.

Interventions: consisted of either sodium fluoride (NaF) or silver diamine fluoride (SDF), as determined by random assignment. In each city, two trained operators conducted the interventions per group. The NaF group received a 5% sodium fluoride varnish (Duraphat Varnish, Colgate-Palmolive, Germany), and the SDF group received a 38% silver diamine fluoride solution (Step 1 Riva Star - Southern Dental Industries (SDI) Limited, Australia), following the manufacturers' guidelines. Prior to treatment, parents and children were informed about possible staining of teeth and soft tissues, without disclosing group assignments.

During the intervention, operators assessed each child's behavior using Frankl's Behavior Rating Scale (Definitely Positive; Positive; Negative; Definitely Negative). Afterward, children self-assessed pain intensity using the Visual Analogue Face Scale, selecting one of five facial expressions (ranging from a smiling face for "Very light pain" to a crying face for "Unbearable pain").

Parents rated their satisfaction with the dental procedure on a 5-point Likert scale adapted from the Treatment Evaluation Inventory (TEI), with options from "Very satisfied" to "Very dissatisfied." At six months, the same intervention was repeated for each child by the same group of operators.

Adverse Effects: One day after the initial intervention and again at the 1-year follow-up, a trained examiner (blinded to the type of intervention) assessed the children for any adverse effects on soft tissues, specifically checking for irritation, inflammation, or pigmentation of the gums or mucous membranes.

Statistical Analysis: Clinical and demographic data, along with assessments of child behavior, pain, and parental satisfaction, were recorded digitally in a secure Microsoft Excel® (2010) database with limited access. The data were organized into a validated dataset and analyzed by an independent statistician using R version 4.3.1, with all tests two-tailed and a significance level of 0.05. Parametric tests were prioritized, but nonparametric methods were used for data that did not meet parametric assumptions, as determined by the Shapiro-Wilk test. Non-normally distributed variables were analyzed using the Mann-Whitney U test.

Participant demographics and clinical characteristics (city, sex, age), as well as oral health practices, adherence, fidelity, child behavior, pain, and parental satisfaction, were summarized using counts and percentages. Inter-examiner reproducibility for caries assessment was measured with a weighted kappa based on ICDAS criteria, maintaining a minimum kappa of 0.7, and intra-examiner reproducibility was assessed using the ICDAS-merged Epi criteria for consistency.

Caries experience (dmfs) was defined by 'decayed/cavity' (d) (ICDAS-merged Extensive caries), 'missing' (m), and 'filled' (f) tooth surfaces (s). Additionally, Initial and Moderate lesions were included in the ICDAS-merged Epi caries experience (ICDAS-merged Epi dmfs). At baseline, the proportion of subjects and the mean number (SD) of tooth surfaces with dmfs and ICDAS-merged Epi dmfs were calculated. Comparisons between children who remained in the study and those who exited early included the mean number (SD) of dmfs surfaces and five assessed oral health behaviors.

For binary outcomes, generalized linear models (GLMs) with a logit link were applied using R's glm function to calculate odds ratios, estimating the likelihood of new decayed surfaces between intervention and control groups. An odds ratio greater than 1 indicated a higher likelihood of decay in the intervention group, while an odds ratio less than 1 indicated a protective effect.

Chi-square tests assessed differences in child cooperation and parental satisfaction between groups, while adverse effects observed at 1-day and 1-year follow-ups were summarized with descriptive statistics. Both parametric and nonparametric tests were applied as appropriate to detect significant differences between treatment groups at each follow-up, with α = 0.05 set as the threshold for statistical significance.

ELIGIBILITY:
Inclusion Criteria:

* 3-4-year-old children (from Bogotá/Cartagena)
* Informed consent signed.
* Self-reported good general health (parents)

Exclusion criteria:

* Intention to move in the next 12 months
* Systemic disease, physical/mental disability
* Regularly medication intake
* Non-cooperative children

Ages: 3 Years to 4 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 814 (Actual)
Dates: Start 2022-08-22 (Actual); Primary Completion 2023-04-30 (Actual); Study Completion 2024-04-30 (Actual)

PRIMARY OUTCOMES:
one-year proportion of children with new cavities and mean number of new cavities (preventive effect) | 12 months
  The one-year proportion of children with new cavities and the mean number of new cavities reflect the preventive effect of the intervention. These measures help assess how effective the dental treatments (NaF or SDF) were in preventing the development of new carious lesions over the course of the year.
  Proportion of children with new cavities: This refers to the percentage of children who developed new carious lesions (cavities) after one year, compared to the total number of children initially assessed. A lower proportion suggests that the intervention was effective in preventing new cavities.
  Mean number of new cavities: This refers to the average number of new cavities per child in the intervention group. A lower mean number of new cavities indicates a stronger preventive effect, showing that fewer cavities developed over the year in the group that received the intervention.
one-year proportion of children with inactive cavities and mean number of inactive cavities (arresting effect) | 12 months
  The one-year proportion of children with inactive cavities and the mean number of inactive cavities reflect the "arresting effect" of the intervention. These metrics assess how effective the treatment (NaF or SDF) was in halting the progression of existing carious lesions, potentially leading to arrested or inactive cavities.
  Proportion of children with inactive cavities: This refers to the percentage of children who had cavities that became inactive (arrested) after one year. Inactive cavities are characterized by hard, shiny surfaces, indicating that the decay process has stopped. A higher proportion suggests that the intervention was effective in arresting caries progression.
  Mean number of inactive cavities: This refers to the average number of cavities per child that became inactive over the course of one year. A higher mean number of inactive cavities indicates that a greater number of cavities were successfully arrested in the intervention group.

SECONDARY OUTCOMES:
Feasibility at one year, in terms of adherence (number of participants recruited and retained) | 12 months
  Feasibility at one year, in terms of adherence, is measured by tracking the number of participants initially recruited and those who remained in the study throughout the year. This involves comparing the baseline number of enrolled participants with those who completed the 1-year follow-up. High retention rates indicate good adherence and suggest that the study's design, intervention, and follow-up procedures were feasible and acceptable to participants.
Feasibility at one year, in terms of fidelity (number of participants not receiving a different intervention) | 12 months
  Feasibility at one year, in terms of fidelity, refers to the extent to which participants consistently received the intervention to which they were originally assigned, without attending to a different intervention. This is assessed by tracking the number of participants who completed the study without receiving an intervention such as filling. High fidelity ensures that the results of the study can be attributed to the specific intervention, rather than variations in treatment.
Number of participants with adverse oral soft tissue effects (one day after the first intervention and after one year) | 1 day and 12 months
  The number of participants with adverse oral soft tissue effects one day after the first intervention refers to the count of children who exhibited any negative reactions in the oral soft tissues (such as irritation, inflammation, or pigmentation) following the initial application of NaF or SDF. These effects were assessed by a trained examiner who was blinded to the type of intervention. Adverse effects observed one day after treatment help evaluate the immediate safety of the interventions and provide insight into potential short-term side effects.
Satisfaction/acceptance of parents' children with caries care after the first intervention | 12 months
  Satisfaction and acceptance of parents and children with caries care after the first intervention were measured using a self-assessment scale, specifically a 5-point Likert scale. Parents were asked, "How satisfied do you feel with the dental procedure used by the dentist on your child?" The response options were: 5-Very satisfied; 4-Satisfied; 3-Neutral; 2-Dissatisfied; 1-Very dissatisfied. The assessment considered factors such as the effectiveness of the treatment, the comfort level of the child during the procedure, and the overall experience. High levels of satisfaction and acceptance indicated that the intervention was well-received, which suggested that parents were likely to support continued treatment and remain engaged in the study.
Child's self-reported pain | After the dental intervention
  Child's self-reported pain refers to the level of discomfort or pain experienced by the child after the dental intervention, as reported by the child themselves. In the study, children assessed their pain intensity using a Visual Analogue Face Scale. This scale includes five facial expressions ranging from a smiling face indicating "very light pain" to a crying face indicating "unbearable pain." The child pointed the face that best represented their level of pain. This self-report tool helps gauge the child's pain experience during the dental procedure and provides insight into the perceived comfort or discomfort associated with the intervention.
Child's behaviour (during the procedure) | During the dental intervention
  Child's behavior during the procedure refers to how the child responded emotionally and physically during the dental treatment. This was assessed by the operator using Frankl's Behaviour Rating Scale, which categorizes the child's behavior into four levels from "Definitely Positive" to "Definitely Negative" were the child was highly uncooperative, distressed, or fearful, making it difficult to perform the procedure. This assessment helps evaluate the child's emotional response to the treatment and provides insight into how well the child tolerated the procedure.

CONTACTS AND LOCATIONS:
Overall Officials: Stefania Martignon, PhD, Principal Investigator — Universidad El Bosq
Locations (2):
- Colombia (2):
  - Universidad El Bosque, Bogotá, Bogotá DC
  - Corporación Universitaria Rafael Núñez, Cartagena, Departamento de Bolívar

IPD SHARING:
Plan to Share IPD: No
Plan to Share papers